CLINICAL TRIAL: NCT06016166
Title: The Effects of Eye Mask on Increasing the Sleep Quality and Tear Layer Function in Patients With Dry Eye Disease
Brief Title: Eye Mask on Sleep Quality and Tear Layer Function in Patients With Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamideh Sabbaghi (Other)
Responsible Party: Sponsor-Investigator, Hamideh Sabbaghi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: IR.SBMU.RETECH.REC.1402.099
Record Dates: First submitted 2023-08-15; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye mask users (Experimental): The eyes of the patients will be defined as the intervention
  Interventions: Device: Eye mask
- Non eye mask users (No Intervention): The eyes of the patients will be defined as the controls

INTERVENTIONS:
Device: Eye mask — The 3D eye mask with the ability to adjust for different faces and eliminate light
  Arms: Eye mask users

SUMMARY:
This randomized clinical trial (RCT) was aimed to determine the effects of eye masking on sleep quality and tear layer function in patients with dry eye disease. In this regard, a total of 34 patients with dry eye disease aged between 20 to 35 years old will be participated. They will be randomly divided into case and control (n=17) groups. Patients in the case group will be instructed to wear the eye mask as long as two weeks and the controls will be recommended to not wear it at the same time. Afterwards, the eye mask application will be cross- over for the next 2 hours between the two groups. Tear layer will be investigated in baseline and repeated in both follow- ups of weeks 2 and 4, either quantitatively and qualitatively, by using Schirmer and TBUT tests. Furthermore, the sleep quality will be checked by the PSQI test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dry eye disease according to the OSDI test

Exclusion Criteria:

* Patients with eye disease except dry eye
* Patients using systemic and ophthalmic drugs
* Patients using sleeping and sedative pills

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The effect of using eye mask on tear layer functions between baseline and follow- ups of weeks 2 and 4 in patients with dry eye | between baseline and follow- ups of weeks 2 and 4
  Tear film function is measured quantitatively and qualitatively by the Schirmer (based on millimeters) and TBUT ( based on seconds) test
The effect of using eye mask on sleep quality between baseline and follow- ups of weeks 2 and 4 in patients with dry eye | between baseline and follow- ups of weeks 2 and 4
  Sleep quality is measured by PSQI test based on the obtained score

CONTACTS AND LOCATIONS:
Locations (1):
- Hamideh Sabbaghi, Tehran, Iran